CLINICAL TRIAL: NCT01055886
Title: Supplemental Nicotine Administration for Smoking Cessation in PTSD
Brief Title: Supplemental Nicotine Administration for Smoking Cessation in Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00013158
Record Dates: First submitted 2010-01-24; First posted 2010-01-26 (Estimated); Results first posted 2014-12-15 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2013-11

CONDITIONS: Smoking Cessation
Keywords: PTSD; smoking cessation; nicotine patch
MeSH Terms: conditions — Smoking Cessation; Stress Disorders, Post-Traumatic | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicotine Patch (Active Comparator): Nicotine patch given pre-quit attempt at weeks 4 through 6
  Interventions: Drug: nicotine patch
- placebo patch (Placebo Comparator): placebo patch given pre-quit from weeks 4 through 6
  Interventions: Drug: placebo patch

INTERVENTIONS:
Drug: nicotine patch — Nicotine patch, 7-21 mg.
  Other Names: Nicoderm, Habitrol
  Arms: Nicotine Patch
Drug: placebo patch — placebo patch used from weeks 4-6
  Arms: placebo patch

SUMMARY:
The investigators propose to evaluate the relationship between PTSD, mood, craving and withdrawal symptoms and factors associated with relapse in the context of a randomized clinical smoking cessation trial. The use of supplemental nicotine administration (SNA) during a "pre-treatment" phase before a targeted quit date is an innovative development in smoking cessation, and may be helpful in treating smokers with PTSD. The use of SNA during ad lib smoking for smokers with PTSD is predicted to reduce both the physiological and emotional dependence on inhaled nicotine, thereby increasing the odds of successful smoking cessation.

Smokers with PTSD will be randomly assigned to 1 of 2 pre-cessation patch therapy conditions (active patch versus placebo patch) for 2 weeks before a target quit-smoking date. All participants will receive brief cognitive-behavioral therapy (CBT) and will begin standard nicotine replacement therapy on their quit day. PTSD symptoms, mood, smoking craving and withdrawal symptoms will be evaluated using electronic diary assessment for one week prior to the pre-cessation period, during the 2-week pre-cessation period, and 6 weeks post quit date. The study is designed to address the following aims:

Specific Aim 1: To examine the effects of SNA on PTSD symptoms, mood, craving and withdrawal through electronic diary assessment.

Hypothesis 1.1. SNA will decrease craving for cigarettes during the 2 week pretreatment period as compared to the placebo patch condition.

Hypothesis 1.2. SNA will decrease the perceived improvement in mood and PTSD symptoms associated with smoking behavior.

Hypothesis 1.3. SNA during the pre-cessation period will result in a reduction of withdrawal symptoms following the quit-date.

Specific Aim 2: To evaluate the effect of SNA on quit rates among smokers with PTSD.

Hypothesis 2. SNA during the pre-cessation period will result in improved quit rates Specific Aim 3: To investigate potential predictors of relapse including PTSD symptom severity, mood, anxiety sensitivity, distress tolerance, and self-efficacy.

Hypothesis 3.1 - 3.5 Increased PTSD symptom severity, increased baseline negative affect, increased anxiety sensitivity, decreased distress tolerance, and lower self-efficacy each will independently be associated with shorter abstinence from smoking.

ELIGIBILITY:
Inclusion Criteria:

* between ages of 18 and 70
* smoker who has smoked 10 or more cigarettes per day during past year
* current PTSD
* English speaker
* study physician clearance

Exclusion Criteria:

* organic mental disorder, schizophrenia, current manic syndrome, lifetime but not current PTSD, or current substance abuse/dependence
* pregnancy
* unstable medications
* myocardial infarction in past 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2009-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick S. Calhoun, Ph.D., Principal Investigator — VA Medical Center; Duke University Medical Center
Locations (1):
- VA Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 110 participants signed consent. 41 were excluded: 25 didn't have current PTSD, 7 had contraindicated other psychiatric disorder, 6 didn't meet smoking criteria, 1 was not willing to quit smoking, 1 didn't want to participate after signing consent, and 1 left before completing screen. Another 4 were lost to contact or w/d before randomization.
Period: Overall Study
Arm/Group | Nicotine Patch | Placebo Patch
Started | 33 | 32
Reached Pre-quit Period | 30 (2 withdrawals, 1 lost to contact) | 31 (1 lost to contact)
Completed | 28 (This includes those who completed all sessions and those with w/d post quit (missing = smoking).) | 21 (This includes those who completed all sessions and those with w/d post quit (missing = smoking).)
Not Completed | 5 | 11
Not completed — Withdrawal by Subject | 4 | 9
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by PI | 0 | 1

BASELINE CHARACTERISTICS:
Population: 65 participants were randomized and began study procedures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotine Patch | Placebo Patch | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.15 (10.57) | 42.69 (7.81) | 41.91 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 14 | 15 | 29
Region of Enrollment [Number; unit: participants]
  United States | 33 | 32 | 65

OUTCOME MEASURES:

1. Primary Outcome: Participants Self-reporting Abstinence During 6 Weeks Post Quit
Description: In the 6 week post-quit period, participants completed ecological momentary assessment (EMA), or diary, ratings of their smoking behavior. This outcome reflects the number of participants who reported not relapsing (i.e., smoking 7 days in a row) during the 6 weeks post-quit.
Time Frame: 6 weeks post-quit (from quit date to Session 12); evaluated weekly from Session 7 to Session 12
Population: 37 participants completed the ecological momentary assessment (EMA; diary) ratings during the post-quit period.
Measure: Number; unit: participants
Arm/Group | Nicotine Patch | Placebo Patch
Number analyzed (Participants) | 20 | 17
participants | 16 | 13

2. Secondary Outcome: Abstinence as Measured by Exhaled Carbon Monoxide (CO)
Description: This outcome reflects the number of participants whose exhaled carbon monoxide (CO; a measure of smoking) indicated abstinence (i.e., 6 parts per million or less) at Session 12, which occurred six weeks post-quit.
Time Frame: Session 12, 6 weeks post-quit
Population: Data was available on 30 participants who attended Session 12.
Measure: Number; unit: participants
Arm/Group | Nicotine Patch | Placebo Patch
Number analyzed (Participants) | 15 | 15
participants | 8 | 7

3. Other Pre Specified Outcome: Diary Ratings of Cravings
Description: Participants provided (through ecological momentary assessment) ratings of their smoking craving. This outcome reflects differences between ad lib (or typical) smoking craving compared to smoking craving reported during the pre-quit period. Craving was reported from a single item "Please indicate your desire/craving to smoke," and answers were provided in a 5-point Likert scale where 1=no craving and 5=severe craving. Higher scores are presumed to be "worse" because they indicate increased craving, which is likely to lead to non-abstinence.
Time Frame: During pre-quit period; two weeks
Population: 61 participants provided this EMA data during the pre-quit period.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Nicotine Patch | Placebo Patch
Number analyzed (Participants) | 30 | 31
units on a scale
  Ad Lib period | 2.88 (0.14) | 3.11 (0.14)
  Patch pre-treatment period | 2.57 (0.14) | 2.84 (0.14)

ADVERSE EVENTS:
Arm/Group | Nicotine Patch | Placebo Patch
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 19/30 | 15/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Patch (N=30) | Placebo Patch (N=31)
Nausea (Gastrointestinal disorders) | 5 (5) | 5 (5)
Skin irritation at patch placement site (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5)
Vivid dreams or nightmares (Psychiatric disorders) | 6 (6) | 3 (3)
Increased PTSD symptoms (Psychiatric disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Elevated blood pressure (Cardiac disorders) | 0 (0) | 1 (1)
Increased heart rate (self-reported) (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No